CLINICAL TRIAL: NCT05074511
Title: Weight Variations Impacts on the Ankle of the Child
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant. Professor of physical therapy, Department of Physical Therapy for Pediatrics, Delta University for Science and Technology
Other Study IDs: ankle stability
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Ankle Injuries; Risk of Falling; Stability
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy: Children in this group will be healthy category according to CDC (Centers for Disease Control and Prevention) growth chart which ranged from BMI-for-age 5th to 85th percentiles
- overweight: Children in this group will be overweight category according to CDC (Centers for Disease Control and Prevention) growth chart which ranged from BMI-for-age 85th to 95th percentiles .
- obese: Children in this group will be obese category according to CDC chart which ranged from BMI-for-age > 95th percentiles
- underweight: Children in this group will be underweight category according to CDC chart ranged from BMI-for-age < 5th percentiles

SUMMARY:
Obesity is a global health problem. It changes the measurement of the human body and makes a big change to move the body. The increased weight and mass change the way the limbs and whole body generate and react to force Excess fat also interferes with joint-muscle interactions that are important for functional capacity and postural balance The tendency to increase the thickness of the abdomen contributes to anterior movement of the COM of the body. The purpose of the study is to investigate the biomechanical effect of weight on foot stability in children.

ELIGIBILITY:
Inclusion criteria:

* Their age will be ranging from 7 to 9 years.
* All children have normal stature for age percentile according to CDC chart.
* The sample will include both sex and will be divided in to 4 groups according to the CDC (Centers for Disease Control and Prevention) growth charts
* All children are normal &perform all activities of daily living
* They were able to understand and follow verbal commands and instructions included in the testing procedures.

Exclusion criteria:

* All of them could be part of recreational activities in their public schools but no competitive sports. Children who participated in any regular sport activities involving the lower extremities will be excluded.
* None of them had any surgical intervention in the lower extremities.
* None of them had any history of musculoskeletal deformities or neuromuscular disorders.
* They had neither visual, auditory defect.

Ages: 7 Years to 9 Years | Sex: All
Age Groups: Child
Study Population: Two hundred healthy non-athletic children from both sexes will participate in this study.
  They will randomly be recruited from primary school stage.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
risk of falling in static and dynamic situations for each group | assessed immediately after the procedure
  The Biodex Balance System will be used to assess risk of falling
dynamic level of stability for each group | assessed immediately after the procedure
  The Biodex Balance System will be used to assess level of instability
dynamic Postural stability for each group | aassessed immediately after the procedure
  The Biodex Balance System will be used to assess Postural stability
ankle muscles peak and angle specific torque, power and work for each group | assessed immediately after the procedure
  Isokinetic dynamometer will be used to assess ankle muscles (plantarflexors, dorsiflexors, inverstors and evertors muscles). it will be assess the peak and angle specific torque, power and work for those muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt